CLINICAL TRIAL: NCT02203162
Title: Effect of Electronic Cigarette Use on Cough Reflex Sensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-3288
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cough
Keywords: cough; cough reflex sensitivity; electronic cigarette; capsaicin
MeSH Terms: conditions — Cough; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cough reflex sensitivity (Experimental): electronic cigarette exposure
  Interventions: Device: electronic cigarette exposure

INTERVENTIONS:
Device: electronic cigarette exposure — 30 puffs of a disposable electronic cigarette, 30 seconds apart.

SUMMARY:
Although electronic cigarettes (e-cigs) are now widely used, very little information exists regarding the effect of electronic cigarette use (vaping) on the respiratory system. The aim of this study is to evaluate the acute effect of one e-cig vaping session (30 puffs 30 seconds apart) on cough reflex sensitivity in healthy adult nonsmokers.

DETAILED DESCRIPTION:
30 adult nonsmokers will have their cough reflex sensitivity measured at baseline, 15 minutes after an e-cig vaping session, and 24 hours subsequently. One e-cig vaping session will consist of 30 puffs of an e-cg (Blu) 30 seconds apart, which will deliver the approximate nicotine amount delivered by one tobacco cigarette. Cough reflex sensitivity, defined as C5, the concentration of capsaicin inducing 5 or more coughs, is the standard end point of cough challenge studies.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults (age18 years and above)
* nonsmokers

Exclusion Criteria:

* previous smoker
* asthma/other respiratory illness
* acute viral upper respiratory tract infection (common cold) in previous 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Dicpinigaitis, MD, Principal Investigator — Montefiore Medical Center and Albert Einstein College of Medicine
Locations (1):
- Einstein Division/Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
Results of this study have been published in January 2016 as a full manuscript.

REFERENCES:
- [Result] Dicpinigaitis PV, Lee Chang A, Dicpinigaitis AJ, Negassa A. Effect of e-Cigarette Use on Cough Reflex Sensitivity. Chest. 2016 Jan;149(1):161-5. doi: 10.1378/chest.15-0817. Epub 2016 Jan 6. PMID 26291648

RESULTS

PARTICIPANT FLOW:
Groups:
- Electronic Cigarette Exposure: 30 healthy subjects-adult nonsmokers
Period: Overall Study
Arm/Group | Electronic Cigarette Exposure
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: adult nonsmokers
Groups:
- Subjects: all subjects underwent cough challenge testing at baseline and after e-cig exposure
Arm/Group | Subjects
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30
cough reflex sensitivity [Mean (Standard Deviation); unit: log C5] | 0.5 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cough Reflex Sensitivity (Log C5)
Description: Measurement of cough reflex sensitivity to capsaicin (C5) performed 15 minutes and 24 hours after electronic cigarette use session. Changes in cough reflex sensitivity 15 minutes after e-cig use compared to baseline will be assessed. In addition, cough reflex sensitivity 24 hours after e-cig exposure will also be measured, so that duration of any changes noted after 15 minutes can be assessed. Increase in C5 means decrease in cough reflex sensitivity. Capsaicin cough challenge involves subjects breathing in incremental doubling concentrations of aerosolized capsaicin, 1 minute apart, until the concentration of capsaicin (micromolar) inducing 5 or more coughs (C5) is reached.
Time Frame: Baseline, 15 minutes, and 24 hours post-exposure to e-cig.
Measure: Mean (95% Confidence Interval); unit: log C5
Groups:
- Electronic Cigarette Exposure: 30 subjects-healthy adult nonsmokers
Arm/Group | Electronic Cigarette Exposure
Number analyzed (Participants) | 30
log C5
  change after 15 min | -0.29 [-0.43 to -0.15]
  change after 24 hr | 0.24 [0.10 to 0.38]

ADVERSE EVENTS:
Groups:
- Subjects: 30 subjects-adult nonsmokers
Arm/Group | Subjects
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes